CLINICAL TRIAL: NCT00871429
Title: Selected Skin Products for Cancer Patients: A Product Satisfaction Survey
Brief Title: Skin Care for Cancer Patients: A Product Satisfaction Survey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Mario Lacouture MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEL080108
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Skin Toxicity
Keywords: skin toxicity; cancer patients; adverse effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Lindi skin care products — Subjects will then be instructed to apply all three products daily for 1 month.
  The products include: Lindi Skin soothing balm (product A), Lindi Skin face serum (product B, and Lindi Skin face wash (product C).
  Other Names: Lindi Skin soothing balm (product A); Lindi Skin face serum (product B); Lindi Skin face wash (product C)

SUMMARY:
This study is being done because the investigators would like to evaluate product satisfaction of three test products (product A, product B, product C) that are available at any drug store. This will be done by measuring any changes in the subjects' answers to the Skindex-16 questionnaire at two time points (at screening and baseline visit and at follow-up visit) and by evaluating their responses to the product satisfaction survey that will be given to them by a study coordinator.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate product satisfaction of the following test articles A, B, and C: Lindi Skin soothing balm (product A), Lindi Skin face serum (product B), and Lindi Skin face wash (product C). This will be done by measuring change in Skindex-16 questionnaire at two time points (baseline and follow-up visits) and by evaluating responses to the investigator administered product satisfaction survey.

The secondary objective of this study is to see if there is any correlation between product satisfaction and grade of skin toxicity based on NCI-CTCAE v.3.0 scale.

Participants in this study will be patients seen at the Northwestern University SERIES clinic or Lurie Cancer Center who are receiving chemotherapeutic and or radiation treatments. Subjects who choose to participate complete a Skindex16 questionnaire, and will after consenting to participate, be given all three test articles A, B, and C to use daily for one month. (These test articles are currently marketed products classified by the FDA as cosmetics).

At the return visit, 1 month after baseline visit, the participant will be asked to return the test articles and complete an investigator administered product satisfaction questionnaire for each test article used. 100 participants will be surveyed. Subjects will be telephoned to check for product compliance after 1 week and 2 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years of age.
* Subjects who have the willingness and ability to understand and provide informed consent to participate in the study and are able to communicate with the investigator.
* Subjects who are seen in the SERIES clinic or Lurie Cancer Center and who are receiving chemotherapy and/or radiation treatment for malignancy
* Subjects who have grade <2 skin toxicity based on NCI-CTCAE v3.0 scale.
* Subjects who are routine cosmetics users

Exclusion Criteria:

* Under 18 years of age.
* Known allergy to any of the ingredients in the assigned products (Appendix C).
* Subjects who have grade 2,3,4 skin toxicity based on NCI-CTCAE v3.0 scale.
* Subjects who are pregnant, breast feeding, or those who are planning on becoming pregnant during test period.
* Subjects who use multiple topical agents on study areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Lacouture, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Haley AC, Calahan C, Gandhi M, West DP, Rademaker A, Lacouture ME. Skin care management in cancer patients: an evaluation of quality of life and tolerability. Support Care Cancer. 2011 Apr;19(4):545-54. doi: 10.1007/s00520-010-0851-8. Epub 2010 Mar 25. PMID 20336328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this study will be patients seen at the Northwestern University SERIES clinic or Lurie Cancer Center who are receiving chemotherapeutic and or radiation treatments.
Period: Overall Study
Arm/Group | Lindi Skin Participant Flow
Started | 99
Completed | 75
Not Completed | 24
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 17
Not completed — Questionnaire not completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cancer Patients Using Lindi Skin Products
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 99
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Product Satisfaction of the Following Test Articles A, B, and C: Lindi Skin Soothing Balm (Product A), Lindi Skin Face Serum (Product B), and Lindi Skin Face Wash (Product C)
Time Frame: one month of use
Population: the number of participants for analysis was determined per protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lindi Skin Soothing Balm (Product A) | Lindi Skin Face Wash (Product C) | Lindi Skin Face Serum (Product B)
Number analyzed (Participants) | 75 | 75 | 75
Percentage of Participants
  Participant Product Satisfaction: Very Good/Good | 78.67 | 73.68 | 88.31
  Participant Product Satisfaction: OK | 16.00 | 23.68 | 9.09
  Participant Product Satisfaction: Bad/Very Bad | 5.33 | 2.63 | 2.60

2. Secondary Outcome: Percentage of Subjects With Skin Toxicity Grades 0 to 5 Using The NCI Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 at Baseline Visit and 1 Month Follow-up After Using Lindi Products.
Time Frame: one month
Reporting Status: Not Posted
Measure: Number; unit: Percentage of Participants

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were not collected/assessed.
Arm/Group | Lindi Skin Soothing Balm (Product A) | Lindi Skin Face Wash (Product C) | Lindi Skin Face Serum (Product B)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No limitations of the trial identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No